CLINICAL TRIAL: NCT01794559
Title: A Prospective, Double Blind, Randomized, Multicenter Study to Evaluate the Utility, Safety, and Efficacy of Using PEER Interactive to Inform the Prescription of Medications to Patients With a Primary Diagnosis of a Depressive Disorder Versus Treatment as Usual.
Brief Title: Study to Evaluate the Safety and Efficacy of PEER Interactive Versus Treatment as Usual in Subjects With a Primary Diagnosis of Depression
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: No site recruitment due to Covid-19
Sponsor: MYnd Analytics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNSR011
Record Dates: First submitted 2013-02-14; First posted 2013-02-20 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Depressive Disorder
Keywords: Depression, EEG, QEEG, mTBI, PTSD, efficiency, safety, suicidality
MeSH Terms: conditions — Depressive Disorder; Depression; Stress Disorders, Post-Traumatic; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: This study is prospective in nature. Control group subjects will be treated according to treatment as usual. Experimental group physicians will follow the guidance of the subject's PEER Interactive Report. Subjects will be washed out of medications prior to EEG. The wash out period for outpatients is no longer than 14 days. Subjects will be followed for 6 months after baseline, or until the patient has achieved maximum medical improvement (MMI). Subjects will be seen on a routine basis and assessments will be made at each interaction to evaluate the patient's improvement in mental health. Subjects will be closely evaluated for any psychiatric specific adverse events. The investigator is allowed to treat the patient according to best medical judgment, which may include adding or changing medications, seeing the patient more frequently, or other interventions such as the use of sleep aids.
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject is masked as to assignment to Control or Treatment Group.
  The blinded subject acts as the blinded rater in providing the primary outcome measure of the QIDS-SR16
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Informed by PEER Interactive Report (Experimental): The PEER Interactive Report -This study is prospective in nature. For subjects in the experimental group, the treating physician will follow the guidance of the subject's PEER Interactive Report as regards sensitivity to on-label medications and classes of medication.
  The subjects will be washed out of all current medications prior to having an EEG, which is necessary to generate the PEER Interactive Report. The wash out period for outpatients is no longer than 14 days.
  The subjects will be followed for 6 months after the initial treatment, or until the patient has achieved maximum medical improvement (MMI). The patient will be seen on a routine basis and assessments will be made at each interaction to evaluate the patient's improvement in mental health.
  Interventions: Device: PEER Interactive Report
- No Report (No Intervention): This study is prospective in nature. Subjects in the control group will be treated according to treatment as usual and best judgment of the treating physician. PEER Interactive Report is not provided to the investigator. The subjects will be followed for 6 months after the initial treatment, or until the patient has achieved maximum medical improvement (MMI). The patient will be seen on a routine basis and assessments will be made at each interaction to evaluate the patient's improvement in mental health.

INTERVENTIONS:
Device: PEER Interactive Report — The PEER Interactive Report provides information comparing the subject's Quantitative Electroencephalography (QEEG) to a database of outcomes from patients with similar QEEG results, and how they responded to on-label treatments. This report provides a probability of how this subject will respond to treatment based upon a comparison of similar subjects in the database.
  Arms: Informed by PEER Interactive Report

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, controlled study to evaluate the effectiveness of PEER Interactive to inform treatment in subjects with a primary diagnosis of depression with comorbidity of non-psychotic behavioral disorders versus treatment as usual, as determined by the investigator. The primary measurement for improvement of the subjects depression will be a self-evaluation questionnaire, Quick Inventory of Depressive Symptomatology-Self Report 16, but the investigators will also collect information on their clinical global improvement and any reduction in adverse events.

DETAILED DESCRIPTION:
This study is prospective in nature. Subjects in the control group will be treated according to treatment as usual and best judgment of the treating physician. For the experimental group the treating physician will follow the guidance of the subject's PEER Interactive Report as regards sensitivity to on-label medications and classes of medication.

The subjects will be washed out of all current medications prior to having an EEG, which is necessary to generate the PEER Interactive Report. The wash out period for outpatients is no longer than 14 days.

The subjects will be followed for 6 months after the initial treatment, or until the patient has achieved maximum medical improvement (MMI). The patient will be seen on a routine basis and assessments will be made at each interaction to evaluate the patient's improvement in mental health. The subjects will also be closely evaluated to determine if they are experiencing any psychiatric specific adverse events. The investigator is allowed to treat the patient according to their best medical judgment, which may include adding or changing medications, seeing the patient more frequently, or other interventions such as the use of sleep aids.

ELIGIBILITY:
Inclusion Criteria:

* Must speak and read English
* Must be able to provide written informed consent
* A primary diagnosis of a DSM-IV depressive disorder
* Co-morbidities of non-psychotic behavioral disorders, including PTSD and mild Traumatic Brain Injury (mTBI) are eligible to participate.
* Able to stop all medications (wash out) for 5 half-lves of all medication(s) which affect the EEG. Outpatient subjects are eligible if they can be washed out of their medications in 14 days or less.
* Ability to comply with the requirements of the study

Exclusion Criteria:

* Diagnosis of a psychotic disorder
* History of, or current, open head trauma
* Subjects who would not be good candidates to be washed out of their medications, in the opinion of the investigator.
* History of craniotomy, cerebral metastases, cerebrovascular accident, current diagnosis of seizure disorder, bipolar disorder, schizophrenia, schizo-affective disorder, dementia, mental retardation, or major depression with psychotic features, or use of depot neuroleptics in the last 12 months.
* Clinically significant medical illness, including thyroid disorders.
* Participation in any other therapeutic drug study within 60 days preceding inclusion in the study.
* Know pregnancy and/or lactation, or intent to become pregnant during the study.
* Chronic or acute pain requiring prescription medication(s).
* Candidates with any metal, shrapnel or other similar objects in the head that could affect the QEEG
* Candidates that are currently stable and considered to be at maximum medical improvement on current medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1922 (Estimated)
Dates: Start 2013-03-01; Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Reported 16 (QIDS-SR16) | 6 months
  A 16 question self administer survey on the status of the subject's depression. The measurement will be taken until the completion of the study (6 months)or until the subject achieves maximum medical improvement.

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | 6 months
  A CGI for Improvement (CGI-I) and a CGI of Severity (CGI-S) will be measured at each visit during the study or until the subject reaches maximum medical improvement
Concise Health Risk Tracking (CHRT-7SR) | 6 months
  Self reported survey on suicidality will be conducted at each visit until the completion of the study or until the subject reaches maximum medical improvement.
Post traumatic stress disorder checklist - civilian | 6 months
  A 17 question self-reported measure of the Diagnostic and Statistical Manual (DSM)-IV symptoms of PTSD.
Maximum Medical Improvement (MMI) | 6 months
  At what point in time, if ever, does the subject reach their maximum medical improvement.

OTHER OUTCOMES:
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | 6 months
  Noting the frequency and severity of psychiatric specific adverse events to determine if the information provided in the PEER Interactive Report results in providing treatment that was better tolerated than treatment as usual.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Iosifescu, MD, PhD, Principal Investigator — Langone Center, NYU; Michael Metzig, BA, Study Director — MYnd Analytics, Inc.
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data with other researchers.